CLINICAL TRIAL: NCT04089852
Title: Nitrous Oxide for Pain Management During Intrauterine Device Insertion in Nulliparous Adolescent Women
Brief Title: Nitrous Oxide for Pain Management During IUD Insertion in Nulliparous Adolescent Women
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Not able to perform intervention in current physical clinic location
Sponsor: Boston Children's Hospital (Other)
Collaborators: Praxair Distribution, Inc. (Unknown)
Responsible Party: Principal Investigator, Amy DiVasta, MD, Associate Professor of Pediatrics, Harvard Medical School; Director, Young Women's Health Research; Co-Director, Adolescent Long-Acting Reversible Contraception (LARC) Program; Attending Physician, Division of Adolescent/Young Adult Medicine, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 000000
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Contraceptive Devices; Long-Acting Reversible Contraception; Analgesia; Adolescent Health; Gynecology
MeSH Terms: conditions — Agnosia | interventions — Endothelium-Dependent Relaxing Factors; Inhalation; Oxygen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inhaled nitrous oxide anesthesia (Experimental): Patients will be assigned to a "pre-implementation" (control) group or a "post-implementation" (treatment) group. The first twelve participants will be the control group and the next twelve participants will be the treatment group. The treatment group will receive inhaled N2O/O2. All participants will receive pre-procedural standard of care for IUD insertions, including 400-600 mg ibuprofen orally at least 20 minutes prior to insertion to reduce post-procedure pain. The N2O will be gradually up-titrated to a goal ratio of 70/30 N2O/O2. N2O/O2 will be administered per Boston Children's Hospital (BCH) N2O sedation protocol. Prior to speculum placement, treatment group participants will receive the inhaled gas until minimal sedation is achieved per BCH sedation guidelines, such that the patient is cooperative, oriented, and tranquil. Inhaled N2O will be administered throughout the duration of the procedure.
  Interventions: Drug: Nitrous oxide gas for inhalation
- Inhaled oxygen placebo (Placebo Comparator): Patients will be assigned to a "pre-implementation" (control) group or a "post-implementation" (treatment) group. The first twelve participants will be the control group and the next twelve participants will be the treatment group. The control group will receive inhaled O2 alone. All participants will receive pre-procedural standard of care for IUD insertions, including 400-600 mg ibuprofen orally at least 20 minutes prior to insertion to reduce post-procedure pain. Control group participants will receive 100% O2 for two minutes prior to speculum placement. Inhaled oxygen will be administered throughout the duration of the procedure.
  Interventions: Drug: Oxygen Gas for Inhalation

INTERVENTIONS:
Drug: Nitrous oxide gas for inhalation — All inhaled gases will be administered via nasal mask using a portable nitrous oxide/oxygen (N2O/O2) machine. Environmental safety will be maintained with an N2O scavenger system and Porter Miniature Vacuum System. The treatment group will receive inhaled N2O/O2. The N2O will be gradually up-titrated to a goal ratio of 70/30 N2O/O2 and will be administered as outlined in the treatment arm description.
  Arms: Inhaled nitrous oxide anesthesia
Drug: Oxygen Gas for Inhalation — All inhaled gases will be administered via nasal mask using a portable nitrous oxide/oxygen (N2O/O2) machine. The control group will receive inhaled O2 alone. Control group participants will receive 100% O2 for two minutes prior to speculum placement. Inhaled oxygen will be administered continuously throughout the procedure as outlined in the control arm description.
  Arms: Inhaled oxygen placebo

SUMMARY:
This pilot study aims to assess the feasibility, acceptability, and effectiveness of using nitrous oxide (N2O) sedation for intrauterine device (IUD) insertions for nulliparous adolescent and young adult women in a primary care clinic setting.

DETAILED DESCRIPTION:
The objective of this research study is to learn more about how to make the intrauterine device (IUD) insertion procedure more comfortable. IUDs are highly effective at preventing pregnancy and are also used to treat gynecological conditions such as endometriosis or heavy periods. Unfortunately, many adolescents and young adults do not get an IUD because the insertion procedure can be painful. Currently, there are no medications that successfully reduce pain during IUD insertion for adolescents in the outpatient clinic setting.

We plan to study if nitrous oxide sedation is a feasible strategy for improving the IUD insertion experience for adolescents and young adult women. Although nitrous oxide is already used to manage pain and anxiety in other medical settings (such as for pain during labor or dental procedures), nitrous oxide sedation has not been rigorously studied for IUD insertions in teenagers and young adults.

During phase one of our study ("pre-implementation phase"), study participants will receive current standard of care (ibuprofen) for managing pain during IUD insertions. In phase two ("post-implementation phase"), study participants will receive nitrous oxide sedation in addition to ibuprofen during IUD insertions. We will survey study participants to assess the feasibility, acceptability, and effectiveness of nitrous oxide sedation for IUD insertions in the primary care clinic setting.

This study will help clinicians understand whether nitrous oxide could be a practical and effective way to manage pain and anxiety for adolescents during IUD insertion procedures. Ultimately, we hope this study will lead to increased satisfaction with the IUD insertion procedure and increased use of this highly effective method of contraception among adolescents.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous (no pregnancy of 24 weeks' duration or longer and not currently pregnant)
* adolescent females (14-24 years)

Exclusion Criteria:

* use of opioids, benzodiazepines, or marijuana within the past 24 hours
* failure to meet medical eligibility criteria for an IUD
* medical contraindications to NSAID use
* relative contraindications to N2O administration, including severe pulmonary disease, congenital heart disease, diseases associated with vitamin B12 deficiency, and sickle cell disease

Ages: 14 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Eligibility of female adolescents/young women is based on requirement for female anatomy (i.e., cervix) for IUD insertion. Eligibility is not based on representation of gender identity.
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Pain management satisfaction: | Immediately after intervention/procedure
  Patient satisfaction with their pain management during the procedure as measured on a 5-item Likert scale with 5 categories: Very satisfied, Satisfied, Neutral, Dissatisfied, Very dissatisfied
Anesthetic acceptability: Proportion reporting that inhaled nitrous oxide anesthesia should be available for IUD procedures | Immediately after intervention/procedure
  Proportion reporting that inhaled nitrous oxide anesthesia should be available for IUD (yes, no, not sure) procedures
Procedural satisfaction: VAS | Immediately after intervention/procedure
  Median visual analog scale (VAS) score for procedural pain management satisfaction, with scores ranging from 0 to 100 with 0=completely satisfied to 100= completely dissatisfied

SECONDARY OUTCOMES:
Experience-expectation discrepancy (pain) | Immediately after intervention/procedure
  Proportion reporting reduction in procedural pain compared to anticipated procedural pain as measured by a choice of 3 responses: The procedure hurt LESS than I expected; The procedure hurt THE SAME as I expected; The procedure hurt MORE than I expected
Experience-expectation discrepancy (anxiety) | Immediately after intervention/procedure
  Proportion reporting reduction in procedural anxiety compared to anticipated procedural anxiety, with 3 answer choices: I felt LESS anxious than I expected; I felt THE SAME level of anxiety as I expected; I felt MORE anxious than I expected
Procedural acceptability (self) | Immediately after intervention/procedure
  Proportion reporting that dislike of the procedure would prevent them from getting another IUD in the future (yes, no, maybe)
Procedural acceptability (peers) | Immediately after intervention/procedure
  Proportion reporting willingness to recommend the IUD procedure to a friend, rated on a 100mm sliding scale ranging from 0 (not at all likely) to 100 (absolutely likely)
Procedure-related anxiety rating | Immediately after intervention/procedure
  Median visual analog scale (VAS) score for overall procedure-related anxiety, with scores ranging from 0 to 100 with 0=not at all anxious to 100=the most anxious
Procedural pain rating | Immediately after intervention/procedure
  Procedural pain rating as measured on a 100-mm visual analog scale (VAS) with scores ranging from 0 to 100, where 0= no pain and 100= the worst pain

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No